CLINICAL TRIAL: NCT07317414
Title: A Randomized Clinical Trial Exploring β-alanine as an Adjunct to First-line Immunotherapy in Advanced Hepatocellular Carcinoma
Brief Title: β-alanine in the Treatment of Advanced Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BARO-HCC
Record Dates: First submitted 2025-12-04; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atezolizumab combined with bevacizumab combined with β- alanine (Experimental): Atezolizumab combined with bevacizumab combined with β- alanine
  Interventions: Drug: Atezolizumab combined with bevacizumab combined with β- alanine
- Atezolizumab combined with bevacizumab (Active Comparator): Atezolizumab combined with bevacizumab
  Interventions: Drug: Atezolizumab combined with bevacizumab

INTERVENTIONS:
Drug: Atezolizumab combined with bevacizumab combined with β- alanine — Atezolizumab (Tecentriq®) + Bevacizumab (Avastin®)+β- alanine
  Arms: Atezolizumab combined with bevacizumab combined with β- alanine
Drug: Atezolizumab combined with bevacizumab — Atezolizumab (Tecentriq®) + Bevacizumab (Avastin®)
  Arms: Atezolizumab combined with bevacizumab

SUMMARY:
This study is a prospective, randomized controlled study on nutritional support and metabolic regulation. It assesses the safety, compliance, and improvement of metabolic/physical-related indicators when using β-alanine within the specified dose range as dietary supplementation, in addition to the standard first-line treatment. The anti-tumor efficacy (ORR, PFS, OS) is the exploratory endpoint.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily participated in the study and agreed to sign the written informed consent. They had good compliance, cooperated with the follow-up, and were over 18 years old at the time of signing the informed consent form, with no restrictions on gender.
* Patients diagnosed by imaging and histological examinations as having unresectable, recurrent, locally advanced or metastatic liver cell carcinoma, or meeting the clinical diagnostic criteria for liver cell carcinoma as defined by the American Association for the Study of Liver Diseases (AASLD); BCLC stage C, with no distant metastasis or lymph node metastasis, or BCLC stage B, who are not eligible for therapeutic surgery
* With measurable lesions (according to the RECIST 1.1 standard, non-lymph node lesions have a CT scan long diameter of ≥ 10 mm, and lymph node lesions have a CT scan short diameter of ≥ 15 mm)
* At least 4 weeks prior to the baseline assessment, radical surgery/local treatment was not suitable, or disease progression occurred thereafter. The treatments included lesion resection, ablation, transcatheter arterial chemoembolization, hepatic artery infusion chemotherapy, radiotherapy, etc. All acute toxic effects during local treatment must be ≤ CTCAE5.0 grade 1.
* For patients undergoing non-surgical sterilization or those of childbearing age, a medically approved contraceptive method must be used during the study treatment period and within 3 months after the end of the study treatment; for non-surgical sterilization patients of childbearing age, the serum or urine HCG test must be negative within 7 days before the study enrollment; and they must be non-lactating; For non-surgical sterilization or male patients of childbearing age, they must agree to use a medically approved contraceptive method with their spouses during the study treatment period and within 3 months after the end of the study treatment.
* The functions of the important organs should meet the following requirements: i. Blood test: Absolute neutrophil count 1.5×109/L, platelet count ≥ 50×109/L, hemoglobin ≥ 90g/L; ii. Liver function: Serum total bilirubin ≤ 3×upper limit of normal; Alanine aminotransferase and aspartate aminotransferase ≤ 5×ULN; Serum albumin ≥ 28 g/L; Alkaline phosphatase ≤ 5×ULN; After conventional liver-protective treatment meets the above standards and can be stable for at least 1 week as evaluated by the investigator, it can be enrolled; iii. Kidney function: Serum creatinine ≤ 1.5×ULN, or creatinine clearance rate ≥ 50 mL/min (using the standard Cockcroft-Gault formula), urine test shows urine protein < 2+; For patients whose urine test at baseline shows urine protein ≥ 2+, 24-hour urine collection should be conducted and the 24-hour urine protein quantification < 1g.
* Coagulation function: The international normalized ratio and activated partial thromboplastin time should be ≤ 1.5 × ULN; if the subject is undergoing anticoagulation therapy, as long as the PT and INR are within the range prescribed by the anticoagulant drug, it is acceptable.

Exclusion Criteria:

* Previously diagnosed with fibrotic plate-like hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma and other components through histological/cytological methods;
* Who have previously received local or systemic anti-tumor treatment, or undergone liver transplantation
* Received radiotherapy within 3 weeks prior to the first administration of the drug
* If there has been a history of esophageal or gastric fundus variceal bleeding caused by portal hypertension within 6 months prior to the first administration of the drug, participation in this study is not permitted. If the gastroscopy indicates severe (G3) varices, participation is not allowed.
* Tumor volume > 50% of liver volume; portal vein tumor thrombus (Vp4, tumor thrombus involving the main portal vein, or the tumor mainly affecting the primary branch of the portal vein on the opposite side of the liver lobe, or the primary branches of the bilateral portal veins) and inferior vena cava tumor thrombus. Note: If the tumor thrombus does not completely block the portal vein, and there is still blood flow visible on imaging, the patient can be included in the study.
* Regardless of the severity, for any patient with any signs or history of bleeding predisposition, or for any patient who experienced any bleeding or bleeding-related event of grade ≥ CTCAE 3 within 4 weeks prior to the first administration of the medication
* Severe bleeding tendency or coagulation dysfunction, or currently undergoing thrombolytic therapy; Arterial and venous thromboembolic events occurred within 6 months before the first administration. Implantable venous port or catheter-derived thrombosis, or superficial venous thrombosis, is excluded in cases where thrombosis stabilizes after conventional anticoagulant therapy
* Uncontrollable hypertension, with systolic blood pressure > 150 mmHg or diastolic blood pressure > 90 mmHg after the best medical treatment, history of hypertensive crisis or hypertensive encephalopathy
* Previous history of myocarditis, cardiomyopathy, or malignant arrhythmia; symptomatic congestive heart failure or left ventricular ejection fraction value < 50% on echocardiography. Symptomatic or poorly controlled arrhythmia, including atrial fibrillation or atrial flutter with a ventricular rate greater than 100 beats per minute.
* Patients who have objective evidence of past and current history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, and severe impairment of lung function
* History of gastrointestinal perforation and/or fistula, intestinal obstruction, extensive bowel resection, Crohn's disease, ulcerative colitis or long-term chronic diarrhea within 6 months prior to the first administration of the drug
* Active pulmonary tuberculosis: Those who are currently undergoing anti-tuberculosis treatment or have received anti-tuberculosis treatment within 1 year prior to the first administration.
* The subjects must not have any active autoimmune diseases or a history of autoimmune diseases; the subjects must not have congenital or acquired immune deficiencies, such as HIV-infected individuals, or must not have received live vaccines within 4 weeks prior to the administration of the study medication or during the study period.
* The subjects are undergoing treatment with immunosuppressants, either systemic or local absorbable hormones, with the aim of achieving immunosuppression (dose > 10mg/day of prednisone or other equivalent efficacy hormones), and they have continued to use these medications within the 2 weeks prior to enrollment.
* The subjects had active infections or experienced unexplained fever above 38.5 degrees Celsius during the screening period or before the first administration (in cases where the fever was caused by the tumor, the subjects could be included in the study).
* The researchers believe that these cases should be excluded from this study. For instance, based on the researchers' assessment, the participants have other factors that might cause the study to be prematurely terminated. Such factors include, for example, the need for combined treatment for other serious diseases (including mental illnesses), severe gastric fundal esophageal varices, severe abnormal laboratory test results, and factors related to family or society that could affect the safety of the participants or the collection of data and samples.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2025-12-24 (Estimated); Primary Completion 2028-12-05 (Estimated); Study Completion 2030-12-05 (Estimated)

PRIMARY OUTCOMES:
The Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale | Within 7 days prior to Day 1 of each treatment cycle (each cycle is 21 days).
  Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Scale score (range 0-52); higher scores indicate less fatigue (better outcome).

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: No
Taking into account the protection of patient information, the clinical data will not be made public.